CLINICAL TRIAL: NCT07112521
Title: Evaluating the Efficacy of Home-Based tDCS for Cancer-Related Cognitive Impairment and Its Moderation by Obesity: A Double-Blind Randomized Controlled Trial.
Brief Title: tDCS Intervention in Breast Cancer Survivors With and Without Obesity Reporting Cognitive Impairment
Acronym: LUMINA-brain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Responsible Party: Principal Investigator, Annette Horstmann, Professor, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: LTDK nro7/2025
Record Dates: First submitted 2025-07-02; First posted 2025-08-08 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer Survivor; Obesity, Overweight
Keywords: tdcs; CRCI; breast cancer survivors; obesity; transcranial direct current stimulation; cancer related cognitive impairment
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: Minimization will be applied to allocate participants to the active or sham tDCS group following a 1:1 ratio. The selected prognostic factors include prior chemotherapy (yes/no), menopausal status (pre/post), and obesity (WHtR ≥ 0.54 = living with obesity; WHtR < 0.54 = not living with obesity).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Experimental)
  Interventions: Device: active tDCS
- sham tDCS (Sham Comparator)
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: active tDCS — The anodal electrode will be placed over the left DLPFC (F3), and the cathodal electrode will be placed over the right supraorbital area (FP2). The current will be gradually ramped up to 2mA over 30 seconds, held constant at 2mA for 29 minutes, and then gradually ramped down to 0mA over the final 30 seconds.
  Arms: Active tDCS
Device: sham tDCS — The anodal electrode will be placed over the left DLPFC (F3), and the cathodal electrode will be placed over the right supraorbital area (FP2). The current will be initially ramped up to 2mA over 30 seconds and immediately ramped back down to 0mA.
  Arms: sham tDCS

SUMMARY:
The goal of this intervention is to investigate whether transcranial Direct Current Stimulation (tDCS) can alleviate Cancer-Related Cognitive Impairment (CRCI) in breast cancer survivors, as measured by changes in brain structures and cognitive performance. To assess the efficacy of tDCS, the investigators will compare outcomes between participants receiving active stimulation and those receiving sham stimulation (a placebo condition where participants believe they are receiving stimulation, but are not).

Participants will:

* Undergo a baseline MRI session
* Receive either active or sham tDCS for six weeks
* Undergo a follow-up MRI session
* Complete cognitive tests and respond to psychosocial questionnaires before, during, and after the tDCS intervention

DETAILED DESCRIPTION:
Cancer-Related Cognitive Impairment (CRCI) is common among breast cancer (BC) survivors, manifesting as deficits in memory, attention, and processing speed, further affecting their quality of life. CRCI is likely multifactorial, influenced by demographic and genetic factors, neuroinflammation, and neuroplasticity changes. On the one hand, obesity is a known risk factor for BC and a poorer prognosis. On the other hand, it is linked to neuroinflammation and structural brain changes that contribute to cognitive impairment. However, its role in exacerbating CRCI remains unclear. Understanding this relationship is crucial for optimizing cognitive rehabilitation strategies. Transcranial Direct Current Stimulation (tDCS) is a promising neuromodulation technique that enhances neuroplasticity, and its potential for home-based application could improve treatment feasibility. This study aims to (1) evaluate the effectiveness of home-based tDCS in improving cognitive function in BC survivors and (2) examine obesity as a potential moderator of treatment outcomes. The investigators will conduct a double-blind, sham-controlled tDCS intervention over six weeks, collecting cognitive assessments and dietary data before, during, and after the intervention. MRI scans will be acquired pre- and post-intervention to assess structural and functional changes in cognition-related regions.

Participants will complete five phases over seventeen weeks: baseline, intervention (acute schedule), intervention (continuing schedule), short-term follow-up, and long-term follow-up:

* Seven of these seventeen weeks are designated as assessment weeks, during which participants complete cognitive tests and maintain a food diary over 2 different days.
* Assessment weeks are scheduled at baseline, every other week throughout the intervention and short-term follow-up, and once during long-term follow-up.
* Questionnaires on sleep, physical activity, cognition, and quality of life are completed once per phase.
* tDCS sessions follow a structured schedule, occurring five times per week during the first three weeks and three times per week during the last three weeks.
* MRI scans are performed at baseline and long-term follow-up.

Cognitive assessment includes three cognitive tests representing three domains known to be impaired following breast cancer (Small et al., 2019):

1. Short-term episodic memory, using the Dot Memory task: a 5x5 grid will be shown on the screen with three cells containing red dots. The grid and dots remained on the screen for 3 seconds, and participants were told to remember which boxes contained the red dots. Then, in a distractor task, participants had to touch all the F's on a screen of E's and F's that is presented for 8 seconds. Finally, participants will be instructed to touch the three boxes that contain the red dots on an empty grid. They will perform the task for 12 trials, taking a 15-second break every 4 trials.
2. Speed processing using the Symbol Search task: Three pairs of symbols will be displayed at the top of the screen. Participants will be instructed to find a pair of matching symbols as quickly as possible from two choices at the bottom of the screen. They will perform the task for 60 trials, taking a 15-second break every 20 trials.
3. Attention, using the Card Matching task: Participants will be presented with images of three playing cards in a row and asked to indicate whether the first and third cards are identical. The cards will then shift one place to the left and a new card will be introduced in the third position. After this practice, the first two cards will be flipped so that the faces are not visible and participants will have to recall the card value in the series that transitions to the first card spot in order to match the card value in the third spot which is visible to the participant. They will perform the task for 60 trials, taking a 15-second break every 20 trials.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Over 18 years old
* Diagnosed with primary adult-onset breast cancer within the last 5 years
* Completed all active cancer treatments at least 3 months prior to study participation
* Capable of fulfilling study requirements, including having internet access.
* Fluent in either Finnish or English
* Have normal or corrected vision and hearing
* Right-handed (based on the Edinburgh Handedness Inventory score; Oldfield, 1971)

Exclusion Criteria:

* Have received primary cancer treatment (chemotherapy, radiotherapy, immunotherapy, or surgery) within the last 3 months
* Have a history of childhood-onset cancer
* Present with acute eczema on the scalp
* Diagnosed with dementia, Alzheimer's disease, multiple sclerosis, or - Parkinson's disease
* Have experienced unconsciousness for more than five minutes due to a head/brain injury within the last 10 years
* Have a history of stroke or transient ischemic attack
* Suffer from claustrophobia
* Are pregnant or breastfeeding
* Have any of the following medical implants or devices: cardiac implantable electronic devices, metallic intraocular foreign bodies, neurostimulation systems, cochlear/ear implants, drug infusion pumps, catheters with metal components, metallic fragments (e.g., bullets), cerebral aneurysm clips, magnetic dental implants, tissue expanders, artificial limbs, non-removable piercings, or face tattoos.
* Weight exceeding 250 kg (the MRI table weight limit) or they are unable to fit within the 70 cm diameter bore of the MRI machine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Attention at post-intervention | From baseline to the end of the intervention at 6 weeks
  Performance in the Matching Cards task under active tDCS compared to sham: the mean number of correct trials.
Short-term episodic memory at post-intervention | From baseline to the end of the intervention at 6 weeks
  Performance in the dot memory task under active tDCS compared to sham: the mean Euclidean distance score.
  The mean Euclidean distance score reflects the distance between the original red dot locations and the recalled locations.
Processing speed at post-intervention | From baseline to the end of the intervention at 6 weeks
  Performance in Symbol Search task under active tDCS compared to sham: prompt-level median response latency for correct trials.

SECONDARY OUTCOMES:
Attention at short-term follow-up | From baseline to 3 weeks after the end of the intervention
  Performance in the Matching Cards task under active tDCS compared to sham: the mean number of correct trials.
Short-term episodic memory at short-term follow-up | From baseline to 3 weeks after the end of the intervention
  Performance in the dot memory task under active tDCS compared to sham: the mean Euclidean distance score.
  The mean Euclidean distance score reflects the distance between the original red dot locations and the recalled locations.
Processing speed at short-term follow-up | From baseline to 3 weeks after the end of the intervention
  Performance in Symbol Search task under active tDCS compared to sham: prompt-level median response latency for correct trials.
Attention at long-term follow-up | From baseline to 9 weeks after the end of the intervention
  Performance in the Matching Cards task under active tDCS compared to sham: the mean number of correct trials.
Short-term episodic memory at long-term follow-up | From baseline to 9 weeks after the end of the intervention
  Performance in the dot memory task under active tDCS compared to sham: the mean Euclidean distance score.
  The mean Euclidean distance score reflects the distance between the original red dot locations and the recalled locations.
Processing speed at long-term follow-up | From baseline to 9 weeks after the end of the intervention
  Performance in Symbol Search task under active tDCS compared to sham: prompt-level median response latency for correct trials.
Gray matter changes at long-term follow-up | From baseline to 9 weeks after the end of the intervention
  Volume of gray matter under active tDCS compared to sham.
Gray matter changes at long-term follow-up | From baseline to 9 weeks after the end of the intervention
  Thickness of gray matter under active tDCS compared to sham.
White matter changes at long-term follow-up | From baseline to 9 weeks after the end of the intervention
  Neurite density index under active tDCS compared to sham.
White matter changes at long-term follow-up | From baseline to 9 weeks after the end of the intervention
  Orientation dispersion index under active tDCS compared to sham.
White matter changes at long-term follow-up | From baseline to 9 weeks after the end of the intervention
  Free-water fraction under active tDCS compared to sham.
Functional connectivity strength measured by Fisher-transformed bivariate correlation coefficients changes at long-term follow-up | From baseline to 9 weeks after the end of the intervention
  ROI-to-ROI functional connectivity as measured by resting-state fMRI under active tDCS compared to sham.
Functional connectivity strength measured by Fisher-transformed bivariate correlation coefficients changes at long-term follow-up | From baseline to 9 weeks after the end of the intervention
  Seed-based functional connectivity as measured by resting-state fMRI under active tDCS compared to sham.

OTHER OUTCOMES:
Dynamics of attention skills throughout the intervention | From baseline to week 1-3-5 during the the intervention
  Performance in the Matching Cards task under active tDCS compared to sham: the mean number of correct trials from each prompted assessment.
Dynamics of short-term episodic memory skills throughout the intervention | From baseline to week 1-3-5 during the the intervention
  Performance in the dot memory task under active tDCS compared to sham: the mean Euclidean distance score from each prompted assessment.
Dynamics of processing speed skills throughout the intervention | From baseline to week 1-3-5 during the the intervention
  Performance in Symbol Search task under active tDCS compared to sham: the mean of the prompt-level median response latency for correct trials.
Depression and anxiety score at post-intervention | From baseline to the end of treatment at 6 weeks
  HADS score under active tDCS compared to sham.
Depression and anxiety score at short-term follow-up | From baseline to 3 weeks after the end of the intervention
  HADS score under active tDCS compared to sham.
Depression and anxiety score at long-term follow-up | From baseline to 9 weeks after the end of the intervention
  HADS score under active tDCS compared to sham.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology, Faculty of Medicine, University of Helsinki, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: Undecided